CLINICAL TRIAL: NCT02135965
Title: Testing Potential Synergistic Effects of Albuterol and Caffeine on Metabolic Rate.
Acronym: CALM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PBRC 28026
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Albuterol; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Albuterol 2mg (Experimental): 2 mg of Albuterol is in a pill form or placebo
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Albuterol 4mg (Experimental): 4mg of Albuterol or placebo is given in pill form
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Caffeine 100mg (Experimental): 100mg of Caffeine or placebo is given in a pill form.
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Caffeine 200mg (Experimental): 200mg of Caffeine or placebo is given in a pill form
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Albuterol 2mg & Caffeine 100mg (Experimental): 100mg of Caffeine in combination with Albuterol 2mg or placebo is given in a pill form.
  Interventions: Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Albuterol 2mg and Caffeine 200mg (Experimental): 200mg of Caffeine in combination with Albuterol 2mg or placebo is given in a pill form.
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Albuterol 4mg and Caffeine 100mg (Experimental): 100mg of Caffeine in combination with Albuterol 4mg or placebo is given in a pill form.
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg
- Albuterol 4mg and Caffeine 200mg (Experimental): 200mg of Caffeine in combination with Albuterol 4mg or placebo is given in a pill form.
  Interventions: Drug: 2mg of Albuterol; Drug: 4mg of Albuterol; Drug: 100mg of Caffeine; Drug: 200mg of Caffeine; Drug: Albuterol 2mg & Caffeine 100mg; Drug: Albuterol 2mg and Caffeine 200mg; Drug: Albuterol 4mg and Caffeine 100mg; Drug: Albuterol 4mg and Caffeine 200mg

INTERVENTIONS:
Drug: 2mg of Albuterol — 2mg of Albuterol on metabolic rate
  Other Names: Albuterol
  Arms: Albuterol 2mg; Albuterol 2mg and Caffeine 200mg; Albuterol 4mg; Albuterol 4mg and Caffeine 100mg; Albuterol 4mg and Caffeine 200mg; Caffeine 100mg; Caffeine 200mg
Drug: 4mg of Albuterol — 4mg of Albuterol on metabolic rate
  Other Names: Albuterol
Drug: 100mg of Caffeine — 100mg of caffeine on metabolic rate
  Other Names: Caffeine
Drug: 200mg of Caffeine — 200mg of Caffeine on metabolic rate
  Other Names: Caffeine
Drug: Albuterol 2mg & Caffeine 100mg — Albuterol 2mg and 100mg of Caffeine
  Other Names: Caffeine; Albuterol
Drug: Albuterol 2mg and Caffeine 200mg — Albuterol 2mg and Caffeine 200mg on metabolic rate
  Other Names: Albuterol; Caffeine
Drug: Albuterol 4mg and Caffeine 100mg — Albuterol 4mg and Caffeine 100mg on metabolic rate
  Other Names: Albuterol; Caffeine
Drug: Albuterol 4mg and Caffeine 200mg — Albuterol 4mg and Caffeine 200mg on metabolic rate
  Other Names: Albuterol; Caffeine

SUMMARY:
The purpose of this study is to define a ratio of Caffeine and albuterol that gives a synergistic increase in metabolic rate.

DETAILED DESCRIPTION:
The study consists of 2 screening visits and 8 study visits. Screening visit 1: about 1 hour fasting from 9pm the prior night. Height and weight is measured, vital signs taken and questionnaires completed. Women will have a urine pregnancy test. Blood draw for chemistry panel and blood count.

Screening visit 2: about 1 hour, Medical history, physical examination, and electrocardiogram (a heart tracing).

Visit 1-8 about 4 hours each. 8 separate occasions, with about 7 days between each visit. ON each visit, blood pressure, pulse and temperature is recorded. A resting metabolic rate (RMR) is measured. After a baseline measurement of about 30 minutes of breathing is taken , a pill will be swallow and metabolism(measured by breathing with a clear plastic hood over the upper body to measure metabolic rate ( the oxygen inhaled and the carbon dioxide exhaled).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between the ages of 18 to 50 years, inclusive.
* Have a body mass index between 19 and 40 kg/M2 ( a number calculated from your height and weight), inclusive.

Exclusion Criteria:

* Female who is pregnant or nursing.
* Woman of childbearing potential and do not agree to use an effective method of contraception during the trial. Acceptable methods include abstinence, barrier methods, intrauterine devices, and hormonal methods of contraception.
* A smoker or use nicotine.
* Take regular medication other than birth control pills.
* Use medications known to alter metabolic rate (some asthma medications).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
A change is being assessed for the combination of Albuterol and Caffeine on Metabolic rate. | Participants will be followed at Baseline and the duration of the study, an expected average of 10 weeks.
  The order of which 8 combinations will be determined randomly (like flipping a coin) and neither the participant nor the study personnel will know what is in the pills. The identity of the pills can be determined by breaking the code in the case of an emergency. 1. Albuterol 2mg; 2. Albuterol 4mg; 3. Caffeine 100mg; 4. Caffeine 200mg; 5. Albuterol 2mg and Caffeine 100mg; 6. Albuterol 2mg and Caffeine 200mg; 7. Albuterol 4mg and Caffeine 100mg; 8. Albuterol 4mg and Caffeine 200mg. The data will be analyzed by computing the metabolic rate. Metabolic rate is measured by breathing with a clear plastic hood over the upper body to measure the oxygen inhaled and the carbon dioxide exhaled.

SECONDARY OUTCOMES:
Respiratory Quotient (RQ) | Participants will be followed at Baseline and the duration of the study, an expected average of 10 weeks.
  The respiratory quotient (RQ) is calculated from a ratio indicating the relation of the volume of carbon dioxide given off in respiration to that of the oxygen consumed.
Pulse rate | Participants will be followed at Baseline and the duration of the study, an expected average of 10 weeks.
  Pulse is the rate at which the heart beats. The pulse is usually called heart rate, which is the number of times the heart beats each minute.
Blood Pressure | Baseline to 8 time points of dose
  When the heart beats, it contracts and pushes blood through the arteries to the rest of your body. This force creates pressure on the arteries. This is called systolic blood pressure or the top number. A systolic blood pressure or the bottom number indicates the pressure in the arteries when the heart rests between beats.
Temperature | Participants will be followed at Baseline and the duration of the study, an expected average of 10 weeks.
  An oral temperature is when the thermometer is placed in the mouth to measure the body heat.
Safety Assessments (lab, adverse events, physical exams and electrocardiograms) | Participants will be followed at Baseline and the duration of the study, an expected average of 10 weeks.
  Labs, adverse events, physical exams and electrocardiograms (ECG or EKG) are assessed to make sure nothing is out of normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States